CLINICAL TRIAL: NCT06762964
Title: Cardiac and Metabolic Effects of Dapagliflozin in the Failing Fontan Circulation: A Phase II, Prospective, Double-Blind Study
Brief Title: CAMEO-FONTAN -Dapagliflozin in the Failing Fontan Circulation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Luke J. Burchill, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-011044
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Fontan Circulation; Single Ventricle Heart Disease; HFpEF - Heart Failure With Preserved Ejection Fraction
Keywords: Fontan; HFpEF; SGLT2 inhibitors
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Experimental)
  Interventions: Drug: Dapagliflozin tablet
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Tablet

INTERVENTIONS:
Drug: Dapagliflozin tablet — Patient will take a 10mg tablet of Dapagliflozin once daily for 24 weeks
  Arms: Dapagliflozin
Drug: Placebo Tablet — Patient will take 10mg placebo tablet once daily for 24 weeks
  Arms: Placebo

SUMMARY:
The purpose of this research is to determine whether treatment with the study drug dapagliflozin for 6 months affects pulmonary capillary wedge pressure (PCWP) at rest and during exercise in adults with failing Fontan circulation.

ELIGIBILITY:
Inclusion Criteria

Subjects are eligible to be randomized in the study only if all the following inclusion criteria and none of the exclusion criteria apply:

1. Signed informed consent prior to any study specific procedures
2. History of Fontan procedure
3. Male or female subject
4. Age ≥ 18
5. Symptoms of dyspnea (NYHA II-III) with no non-cardiac or ischemia explanation
6. Undergoing clinically indicated cardiac catheterization
7. Elevated pulmonary capillary wedge pressure (PCWP) during exercise (≥20 mmHg) ascertained at Visit 1. Patients that have consented to study procedures but do not meet this invasive criterion will be considered as screen failures and will not be randomized.

Exclusion Criteria

1. Type I diabetes
2. Any of the following medications: Insulin or Pramlintide, Sandostatin, Akeega (abiraterone acetate), Growth Hormone (Somatogrogon-GHLA), Lithium, Chloroquine, Hydroxychloroquine, Thioctic acid (alpha lipoic acid), Empagliflozin or Canagliflozin
3. Recent hospitalization (<30 days) or revascularization (<90 days)
4. Significant valvular heart disease (≥moderate stenosis, >moderate regurgitation)
5. Significant Fontan obstruction with resting SVC-IVC gradient >4 mmHg
6. Primary cardiomyopathy (such as amyloid)
7. Dyspnea due to primary lung disease or myocardial ischemia in the opinion of the investigator
8. Severe anemia (hemoglobin <9 gm/dl)
9. Severe kidney disease (estimated GFR<30) or liver disease
10. Women of childbearing potential not willing to use a medically accepted method of contraception OR who are currently pregnant (confirmed with positive pregnancy test) or breast feeding.
11. History of serious hypersensitivity reaction to dapagliflozin
12. Subjects on dialysis
13. Subjects with severe liver disease with history of decompensation including ascites or encephalopathy or variceal bleeding
14. Single ventricle heart disease without Fontan palliation
15. Those with a history of Fontan takedown

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Pulmonary capillary wedge pressure (PCWP) at rest | Baseline, 24 Months
  Pulmonary Capillary Wedge pressure will be determined by right heart catheterization with expired gas analysis. Right heart catheterization with expired gas analysis will be performed at rest. Pulmonary Capillary Wedge Pressure is measured in millimeters of mercury (mmHg).
Pulmonary capillary wedge pressure with feet elevated | Baseline, 24 Months
  Pulmonary Capillary Wedge pressure will be determined by right heart catheterization with expired gas analysis. Right heart catheterization with expired gas analysis will be performed with feet elevated. Pulmonary Capillary Wedge Pressure is measured in millimeters of mercury (mmHg).
Pulmonary capillary wedge pressure at 20W exercise | Baseline, 24 Months
  Pulmonary Capillary Wedge pressure will be determined by right heart catheterization with expired gas analysis. Right heart catheterization with expired gas analysis will be performed at 20W exercise. Pulmonary Capillary Wedge Pressure is measured in millimeters of mercury (mmHg).

SECONDARY OUTCOMES:
Right atrial pressure at rest | Baseline, 24 Months
  Right atrial pressure at rest will be determined by right heart catheterization with expired gas analysis. Right heart catheterization with expired gas analysis will be performed at rest. Right atrial pressure will be measured in millimeters of mercury (mmHg).
Right atrial pressure with exercise | Baseline, 24 Months
  Right atrial pressure at rest will be determined by right heart catheterization with expired gas analysis. Right heart catheterization with expired gas analysis will be performed with exercise. Right atrial pressure will be measured in millimeters of mercury (mmHg).
Pulmonary artery pressures at rest | Baseline, 24 Months
  Pulmonary artery pressures will be determined by right heart catheterization with expired gas analysis. Pulmonary artery pressures with expired gas analysis will be performed at rest. Pulmonary artery pressures will be measured in millimeters of mercury (mmHg).
Pulmonary artery pressures with exercise | Baseline, 24 Months
  Pulmonary artery pressures will be determined by right heart catheterization with expired gas analysis. Pulmonary artery pressures with expired gas analysis will be performed with exercise. Pulmonary artery pressures will be measured in millimeters of mercury (mmHg).
Cardiac output at rest | Baseline, 24 Months
  Cardiac output measures the amount of blood the heart pumps per minute. It is calculated by Cardiac Output= Oxygen Consumption/(Arterial - Venous Oxygen Content Difference). Cardiac output will be measured in liters per minute (L/min).
Cardiac output with exercise | Baseline, 24 Months
  Cardiac output measures the amount of blood the heart pumps per minute. It is calculated by Cardiac Output= Oxygen Consumption/(Arterial - Venous Oxygen Content Difference). Cardiac output will be measured in liters per minute (L/min).
Peak oxygen consumption (VO2) during exercise | Baseline, 24 Months
  Peak oxygen consumption (VO2) is measured in milliliters of oxygen per minute (mL/min).
Change in plasma volume | Baseline, 24 Months
  Plasma volume will be determined by radiolabeled iodinated albumin (131I, 5-25 μCu) indicator dilution technique (BVA-100 Blood Volume Analyzer, Daxor Corp, NY). Plasma volume will be measured in milliliters (mL).
Change in blood volume | Baseline, 24 Months
  Blood volume will be determined by radiolabeled iodinated albumin (131I, 5-25 μCu) indicator dilution technique (BVA-100 Blood Volume Analyzer, Daxor Corp, NY). Blood volume will be measured in milliliters (mL).
SF-36 quality of life (QOL) | Baseline, 24 Months
  SF-36 quality of life (QOL) questionnaire is a 36-question questionnaire that evaluates a patient's quality of life. The score range is from 0-100, with a higher score reflecting a better quality of life.
Change in fat mass | Baseline, 24 Months
  Fat mass will be determined by Dual Energy X-ray Absorptiometry Scan. Fat mass will be measured in kilograms (kg).
Change in fat free mass | Baseline, 24 Months
  Fat free mass will be determined by Dual Energy X-ray Absorptiometry Scan. Fat free mass will be measured in kilograms (kg).

CONTACTS AND LOCATIONS:
Overall Officials: Luke Burchill, M.B.B.S., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No